CLINICAL TRIAL: NCT05343585
Title: Testing the Validity of an Artificial Intelligence-based Program to Identify Foods and Estimate Food Portion Size Among Adults, a Pilot Study
Brief Title: Validity of an AI-based Program to Identify Foods and Estimate Food Portion Size
Acronym: PortionSizeAI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Chloe, Principal Investigator, Pennington Biomedical Research Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PBRC 2022-011; T32DK064584 (NIH)
Record Dates: First submitted 2022-04-12; First posted 2022-04-25 (Actual); Results first posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Nutrition Assessment
Keywords: Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): * Training and use of Openfit
  * Using the app to estimate food intake from simulated meals in a laboratory at PBRC or LSU (participants will not eat food during the meals)
  * Rating the usability and satisfaction of the app
  Interventions: Device: PortionSize AI

INTERVENTIONS:
Device: PortionSize AI — For this pilot study, using a convenience sample, the investigators will recruit up to 25 adults to use the Nutrition AI technology in Openfit to identify and estimate portion size of foods provided in a laboratory setting at Pennington Biomedical Research Center (PBRC) and/or Louisiana State University (LSU). Laboratory members within the Ingestive Behavioral Laboratory will also test the ability of Nutrition AI to identify foods and to quantify foods provided in the laboratory. Meals will be simulated, and participants will not consume the foods provided.

SUMMARY:
The purpose of this study is to test the accuracy of the Nutrition Artificial Intelligence in the Openfit app during meals in a controlled laboratory setting

DETAILED DESCRIPTION:
For this pilot study, using a convenience sample, the investigators will recruit up to 25 adults to use the Nutrition AI technology in Openfit to identify and estimate portion size of foods plated in a laboratory setting at Pennington Biomedical Research Center (PBRC) and/or Louisiana State University (LSU). Laboratory members within the Ingestive Behavioral Laboratory will also test the ability of Nutrition AI to identify foods and to quantify foods provided in the laboratory. Meals will be simulated, and participants will not consume the foods provided.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Aged 18-62 years
* Self-reported body mass index (BMI) 18.5-50 kg/m2

Exclusion Criteria:

* Any condition or circumstance that could impede study completion
* Unfamiliar with or not able to use an iPhone

Ages: 18 Years to 62 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2022-04-27 (Actual); Primary Completion 2022-06-03 (Actual); Study Completion 2022-06-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chloe P Lozano, PhD, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No
Any identifiers might be removed from the participants identifiable information and after such removal, the information could be used for future research studies or given to another investigator for future research without additional informed consent from the subject or legally authorized representative.

REFERENCES:
- [Derived] Lozano CP, Canty EN, Saha S, Broyles ST, Beyl RA, Apolzan JW, Martin CK. Validity of an Artificial Intelligence-Based Application to Identify Foods and Estimate Energy Intake Among Adults: A Pilot Study. Curr Dev Nutr. 2023 Sep 29;7(11):102009. doi: 10.1016/j.cdnut.2023.102009. eCollection 2023 Nov. PMID 38026571

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental: * Training and use of Openfit
  * Using the app to estimate food intake from simulated meals in a laboratory at PBRC or LSU (participants will not eat food during the meals)
  * Rating the usability and satisfaction of the app
  PortionSize AI: For this pilot study, using a convenience sample, the investigators will recruit up to 25 adults to use the Nutrition AI technology in Openfit to identify and estimate portion size of foods provided and simulated plate waste, and food intake in a laboratory setting at Pennington Biomedical Research Center (PBRC) and/or Louisiana State University (LSU). Laboratory members within the Ingestive Behavioral Laboratory will also test the ability of Nutrition AI to identify foods and to quantify foods provided, plate waste and food intake, in the laboratory. Meals will be simulated, and participants will not consume the foods provided.
Period: Overall Study
Arm/Group | Experimental
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Experimental
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.0 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 17
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 24
Education [Count of Participants; unit: Participants]
  Some College or Bachelor's Degree | 10
  Postgraduate degree | 14
Employment [Count of Participants; unit: Participants]
  Full time | 22
  Part time | 2
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 24.6 (4.1)

OUTCOME MEASURES:

1. Primary Outcome: Identification of Food Plated Using the Openfit Mobile App
Description: Agreement surrounding identification of food and beverages provided compared with known identification, at the item level, and across all items where identification is determined by: 1) Nutrition AI without correction (automated), 2) Nutrition AI with user correction (semi-automated)
  For a food identified through the Nutrition AI to be considered an exact food match, the name of the food identified must match or be a close match to the food served. For example, a fruit cocktail identified as a fruit salad is an acceptable match. Proportions will be used to assess whether the percentage of food items plated that were correctly identified by Nutrition AI is different to the percentage of foods correctly identified by a criterion method (human rater). Descriptive data will also be used to describe the frequency at which food plated was correctly identified for all food items across all participants. In total there was 255 food items tested across all participants.
Time Frame: One study visit of ~2 hours
Measure: Count of Units; unit: Food items
Units Other Than Participants: Food items
Arm/Group | Experimental
Number analyzed (Participants) | 24
Number analyzed (Food items) | 255
Food items
  Food items that were automatically identified as an exact match across all participants. | 118
  Food items that were semi-automatically identified as an exact match across all participants. | 221

2. Primary Outcome: Portion Size Estimation (kcal) of Food Plated Using the Openfit Mobile App
Description: Error between mean estimates of food plated (kcal) and known food plated (kcal), determined by: 1) Nutrition AI without user correction (automated), 2) Nutrition AI with user correction (semi-automated)
  Mean error and Bland-Altman analysis will be performed to determine errors in estimation of food plated from the Nutrition AI compared to estimations from the criterion measure (weighed food).
Time Frame: One study visit of ~2 hours
Measure: Mean (Standard Deviation); unit: kcal
Arm/Group | Experimental
Number analyzed (Participants) | 24
kcal
  Energy of weighed meals. | 577 (150)
  Energy of automated estimates | 826 (490)
  Energy of semi-automated estimates | 769 (445)

3. Primary Outcome: User Satisfaction of the Openfit Mobile App for Recording Food Plated
Description: After completing assessment of food plated, participants will complete a user satisfaction survey (USS). The USS was adapted from a previous version used to assess the usability of a mobile application for dietary assessment. The USS includes five quantitative questions and three open response questions. The quantitative questions will each be scored using a 6-point Likert scale, with 1 being the lowest and worst score, and 6 being the highest and best score.
  Data for each of the five quantitative responses in the USS will be averaged across participants and presented separately as mean (SD). Open responses will be evaluated using qualitative methods to identify common themes.
Time Frame: One study visit of ~2 hours
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental
Number analyzed (Participants) | 24
score on a scale
  How satisfied are you with the app for identifying the food provided? | 4.1 (1.3)
  How satisfied are you with the app for estimating the amount of food provided? | 4.0 (1.5)
  How easy was it to use the app to identify the food provided? | 4.2 (1.4)
  How easy was it to use the app for estimating the amount of food provided? | 4.0 (1.6)
  How much did the training help prepare you for using the app? | 5.5 (0.7)

4. Primary Outcome: Usability of the Openfit Mobile App for Recording Food Plated
Description: Participants will complete the Computer Usability Satisfaction Questionnaire (CSUQ). The CSUQ is frequently used to assess the usability of mobile applications. The CSUQ consists of 19 questions, each scored using a 7-point Likert scale (with 1 being the lowest and best score and 7 being the highest and worst score) and participants will rate satisfaction, usefulness, information quality, and interface quality of the Openfit app. The average of these 19 questions (1 being the best average score and 7 being the worst average score) provides an overall usability score.
Time Frame: One study visit of ~2 hours
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental
Number analyzed (Participants) | 24
score on a scale | 2.4 (0.22)

ADVERSE EVENTS:
Time Frame: Over 1 study visit of approximately 2 hours.
Arm/Group | Experimental
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-08): https://cdn.clinicaltrials.gov/large-docs/85/NCT05343585/Prot_SAP_000.pdf